CLINICAL TRIAL: NCT03702634
Title: Chaplain Family Project Randomized Controlled Trial
Brief Title: Chaplain Family Project Trial
Acronym: CFP-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Regenstrief Institute, Inc. (Other); Indiana University Health (Other)
Responsible Party: Principal Investigator, Alexia M. Torke, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1806775750
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; PTSD; Depression; Communication; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression; Communication; Personal Satisfaction | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Arm 1- Control group Arm 2- Intervention group
Who Masked: Outcomes Assessor
Masking Description: Research staff conducting interviews with study participants will be masked to study group allocation, until all outcome assessments for that participant have been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Usual Care) (No Intervention): Surrogate will receive usual care in the hospital, which could include visits from the unit chaplain or other staff from the spiritual care department.
- Intervention (Experimental): Spiritual Care Assessment and Intervention (SCAI) framework
  Interventions: Behavioral: Spiritual Care Assessment and Intervention (SCAI) framework

INTERVENTIONS:
Behavioral: Spiritual Care Assessment and Intervention (SCAI) framework — The study chaplain will work with the surrogate, using questions in four domains of spiritual care, to assess them and tailor the visit to their specific needs. The study chaplain will then utilize a pre-determined list of spiritual care interventions, and also document observable outcomes that occur at each visit (which are also listed within the SCAI framework).
  Arms: Intervention

SUMMARY:
Our research team has designed a chaplain delivered intervention focused on surrogate decision makers for hospitalized adults in the ICU. In this study, surrogates will complete an enrollment interview with research staff, including the completion of anxiety screening (GAD-7). Based on their score the surrogate will be put into one of two groups, and then randomized to either the control or intervention group. Control group members will receive usual care, while intervention group members will meet with our study chaplain, who will provide the SCAI (Spiritual Care Assessment and Intervention) framework.

DETAILED DESCRIPTION:
Unmet spiritual needs may have at least two negative consequences for surrogates. First, they may have high levels of spiritual distress, an important aspect of the surrogate's well-being. Second, surrogates include their religious and spiritual beliefs when making serious medical decisions . Therefore unmet spiritual needs may have a negative effect on the surrogate's ability to make good decisions for the patient, especially when facing extremely distressful decisions such as whether to continue life sustaining treatment or enroll in hospice.

The specific aims of this proposed study are:

1. To determine the effect of the spiritual care intervention on psychological well-being for family surrogates at 3 months post discharge, including anxiety (primary outcome: GAD-7), depression (PHQ-9), Posttraumatic stress (IES-R), and overall distress.
2. To determine the effect of the spiritual care intervention on spiritual well-being for family surrogates, (FACIT-SP- non-illness) and on religious coping (Brief RCOPE positive and negative).
3. To determine the effects of the spiritual care intervention on other aspects of the surrogates' experience, including satisfaction with spiritual care (Patient Satisfaction Instrument--Chaplaincy) communication (FICS), overall satisfaction with the hospital stay (Picker single item) and decision conflict (DCS).
4. To determine the effect of the intervention on treatment at the end of life (life sustaining treatments and hospice utilization) for patients who die in the hospital.
5. To determine differences in outcomes between the intervention group, who will receive our intervention, and the control group, who will receive the usual care provided by the hospital chaplaincy service.

ELIGIBILITY:
Inclusion Criteria:

Cognitive Requirements

1. Patient is not decisional due to:

   * Intubation (other than surgery- see exclusion criteria below)
   * Sedation
   * Unresponsive
   * otherwise unable to communicate (AMS, dementia, delirium, etc.)

   Decision Support Requirements
2. Patient has a qualified surrogate decision maker

Exclusion Criteria:

* Intubated for surgery and expected to be extubated within 24 hours
* Imminently dying as evidenced by patient notes
* Patient and/or family have a care contract or other restriction due to complicated or volatile situation
* Patient is a prisoner
* Patient is being followed by Adult Protective Services (APS)
* Patient meets cognitive criteria but does not have a qualified surrogate decision maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Change in anxiety from baseline enrollment interview to 6-8 weeks post patient discharge | Assessed at enrollment and again 6-8 weeks after hospital discharge
  GAD-7 (7 item inventory of anxiety)

SECONDARY OUTCOMES:
Change in depression from baseline enrollment interview to 6-8 weeks post patient discharge | Assessed at enrollment and again 6-8 weeks after hospital discharge
  PHQ-9 (9 item inventory of depression)
Presence of post traumatic stress at 6-8 weeks post patient discharge | Assessed 6-8 weeks after hospital discharge
  IES-R (Impact of Events scale- inventory for PTSD)
Change in overall distress from baseline enrollment interview to 6-8 weeks post patient discharge | Assessed at enrollment and again 6-8 weeks after hospital discharge
  Distress thermometer (a 1-10 scale developed by our team to assess distress)

OTHER OUTCOMES:
Change in spiritual well-being at baseline enrollment interview to 6-8 weeks post patient discharge | Assessed at enrollment and again 6-8 weeks after hospital discharge
  FACIT-SP- non-illness scale (a validated scale of spiritual well-being)
Change in religious coping from baseline enrollment interview to 608 weeks post patient discharge | Assessed at enrollment and again 6-8 weeks after hospital discharge
  Brief RCOPE (a validated scale of religious coping)
Satisfaction with spiritual care at 6-8 weeks post patient discharge | Assessed 6-8 weeks after hospital discharge
  Patient Satisfaction Instrument- Chaplaincy (an adaptation of a scale of patient satisfaction to be used with surrogates)
Communication in the hospital at 6-8 weeks post patient discharge | Assessed 6-8 weeks after hospital discharge
  Family Inpatient Communication Survey (FICS) (A validated scale of communication
Overall satisfaction with the hospital stay at 6-8 weeks post patient discharge | Assessed 6-8 weeks after hospital discharge
  Picker single item (1-10)
Presence of decision conflict at 6-8 weeks post patient discharge | Assessed 6-8 weeks after hospital discharge
  Decision Conflict Scale (DCS) (a validated scale of decision conflict that is used to assess decision conflict when a person has made 1 or more major decisions for a patient in the hospital setting)
Effect of the intervention on end of life care for those who die in the hospital | Chart abstraction to review from the date of admission to the hospital up to one year after admission
  Will use comparative statistics to determine any correlations between intervention and EOL care (life sustaining treatments received and hospice enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Alexia M Torke, MD, MS, Principal Investigator — Indiana University, IU Health, Regenstrief Institute
Locations (2):
- United States (2):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torke AM, Varner-Perez SE, Burke ES, Taylor TA, Slaven JE, Kozinski KL, Maiko SM, Pfeffer BJ, Banks SK. Effects of Spiritual Care on Well-Being of Intensive Care Family Surrogates: A Clinical Trial. J Pain Symptom Manage. 2023 Apr;65(4):296-307. doi: 10.1016/j.jpainsymman.2022.12.007. Epub 2022 Dec 14. PMID 36526251